CLINICAL TRIAL: NCT00280358
Title: A Study in Healthy Volunteers to Evaluate Serum and Urine Levels of the Investigational Product Versus Comparator.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dey (Industry)
Responsible Party: Director Clinical Affairs, Dey, LP
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 191-072
Record Dates: First submitted 2006-01-19; First posted 2006-01-23 (Estimated); Last update posted 2008-03-07 (Estimated); Status verified 2008-03

CONDITIONS: Healthy
Keywords: Fluticasone; Formoterol; PK Study; Pharmacokinetics
MeSH Terms: interventions — Fluticasone; Formoterol Fumarate

INTERVENTIONS:
Drug: Fluticasone Propionate
Drug: Formoterol Fumarate

SUMMARY:
The purpose of the study is to obtain initial pharmacokinetic data in healthy patients after dosing a combination of the study medications.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers, BMI 18-29, no current medications

Exclusion Criteria:

* Significant conditions or disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Levels of study medication in blood and urine.

SECONDARY OUTCOMES:
Safety/tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Lenexa, Kansas, United States